CLINICAL TRIAL: NCT03356366
Title: Magnetic Resonance Imaging Study of the Mechanisms Underlying Irreversible Disability in Multiple Sclerosis
Brief Title: MRI Study of the Mechanisms Underlying Irreversible Disability in Multiple Sclerosis
Acronym: SEP-MRI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-52; 2017-A00136-47 (Other: ANSM)
Record Dates: First submitted 2017-11-06; First posted 2017-11-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Principal study (Experimental): Patients pathological process will be assessed using MRI 3T
  Interventions: Other: MRI 3T
- Ancillary study 1 (Experimental): Patients pathological process will be assessed using MRI 1,5T
  Interventions: Other: MRI 1,5T
- Ancillary study 2 (Experimental): Patients pathological process will be assessed using MRI 7T
  Interventions: Other: MRI 7T

INTERVENTIONS:
Other: MRI 3T — Magnetic Resonance Imaging 3 Tesla
  Arms: Principal study
Other: MRI 1,5T — Magnetic Resonance Imaging 1,5 Tesla
  Arms: Ancillary study 1
Other: MRI 7T — Magnetic Resonance Imaging 7 Tesla
  Arms: Ancillary study 2

SUMMARY:
Multiple sclerosis (MS) is the first non-traumatic cause of disability in young people, responsible for physical but also cognitive deficits. MS is an inflammatory demyelinating and degenerative disease of the central nervous system. Recently, MRI technics have demonstrated their sensibility to the different processes involved in MS. Particularly, MRI has evidenced that the pathological process of MS is not restricted to the macroscopic lesions of the white matter but also involves the normal appearing white and grey matter. In the normal appearing brain tissue, demyelination, neuronal suffering and neuronal loss have been evidenced. Moreover, MRI has demonstrated the existence of brain functional reorganization processes that may limit the clinical expression of pathological injuries. Despite these important findings, the pathological underpinnings of irreversible disability are largely unknown. The present project aims to depict the main determinants of physical but also cognitive disability in patients with MS. To do this, a longitudinal study including 70 patients with MS using different MRI markers known to be sensitive to the different pathological aspects of MS will be performed. The relationships between these markers and the progression of disability will be assessed. Identification of the main pathological underpinnings of irreversible disability of MS will provide the most relevant therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Major patient,
* Patient affiliated to a health insurance plan
* Patient having signed free and informed consent after receiving detailed, understandable and honest information,
* Patient with multiple sclerosis according to the criteria of Polman 2010

Exclusion Criteria:

* Patients with the usual contraindications to MRI (pace-maker, agitation, metal splinters, claustrophobia etc.)
* Patients at risk of non-compliance on examination: impaired understanding, confusion, involuntary movements, poor tolerance of prolonged supine
* Patients with known allergy to gadolinium
* Patients with renal insufficiency
* Patients unable to give their consent: disorders of the comprehension, disturbances of vigilance, confusion ...
* Pregnant and breastfeeding woman
* Patients with a history of neurological or psychiatric pathology
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of the Expanded Disability Status Scale (EDSS) value (score from 0 to 20) constituing the actual international reference scale to measure the level of disability caused by parkinson disease | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided